CLINICAL TRIAL: NCT00859300
Title: MAP-IDM: Identification of Molecular Markers of Sudden Death at the Acute Phase of Myocardial Infarction. A Case Control Study
Brief Title: MAP-IDM: Identification of Molecular Markers of Sudden Death at the Acute Phase of Myocardial Infarction
Acronym: MAP-IDM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2007.463
Record Dates: First submitted 2008-03-05; First posted 2009-03-11 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; ventricular fibrillation; sudden death; polymorphism
MeSH Terms: conditions — Myocardial Infarction; Ventricular Fibrillation; Death, Sudden | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 500 patients with ventricular fibrillation at the acute phase of myocardial infarct
  Interventions: Genetic: Blood sample
- 2: 500 patients without ventricular fibrillation at the acute phase of myocardial infarct.
  Interventions: Genetic: Blood sample

INTERVENTIONS:
Genetic: Blood sample — Blood sample Determination of genetic background
  Groups: 1
Genetic: Blood sample — Blood sample Determination of genetic background
  Groups: 2

SUMMARY:
We propose a comparative case-control study on the 2 following groups of patients:

* Cases: 500 patients with ventricular fibrillation at the acute phase of myocardial infarct,
* Controls: 500 patients without ventricular fibrillation at the acute phase of myocardial infarct.

The primary endpoint in this study is the correlation phenotype/genotype of sudden death at the acute phase of myocardial infarct.

The first phase of the study, including patients' recruitment, clinical and biological data collection, will last 82 months. The second phase will concern the genotype/phenotype analysis and the identification of polymorphisms associated with a sudden death risk after a myocardial infarction.

This study will allow a better knowledge of the mechanisms of sudden death and the identification of new risk markers.

DETAILED DESCRIPTION:
The number of sudden death is estimated around 50000 in France. In most cases, these deaths are due to myocardial infarction. This complication occurs, for 70% of cases, at the patient's residence, within 30 minutes following the thoracic pain. Emergency care often comes too late and allows only 2% of the patients having a heart failure to be revitalized.

At equal sex, age and clinical status, patients may or not develop ventricular rhythm disorders. Then, the notions of risk background and genetic disposition should be investigated.

No prospective study has been conducted on a sufficient number of patients yet. Such a study and the recent development of new genetic technologies will help identifying markers of sudden death risk at the acute phase of myocardial infarction.

The study we are implementing will increase knowledge on sudden death mechanisms at the acute phase of myocardial infarction. The analysis of phenotypic/genotypic relations will lead to an identification of new risk markers. Further evaluations of new diagnostic and therapeutic strategies will be possible on the basis of this trial.

Ventricular fibrillation at the acute phase of myocardial infarction follows a polygenic determinism. The genes involved in this electrical trouble are those which lead to the expression of potassic, calcic and sodic channels of ventricular myocytes: KCNQ1, KCNH2, SCN5A, KCNE1, KCNE2, KCNJ2, PRKAG2, RyR2, PKP2, DSP, CASQ2, CACNA1C, and FKBP1B.

An association of a favourable genetic background and ischemia represents a cause for ventricular arrhythmia as a complication of myocardial infarction.

Haplotypes or genes considered as new markers for sudden death risk of ischemic origin will be searched.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to ICU for MI and presenting the following criteria:
* Age > 18
* Group 1 (Case) Patients with cardiac arrest and ventricular fibrillation developed up to 24 h post MI Group 2 (control) Patients with MI (no ventricular fibrillation)
* Written informed consent.

Exclusion Criteria:

* No written informed consent
* Known Medical History of cardiomyopathy, including acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases: 500 patients with ventricular fibrillation at the acute phase of myocardial infarct, Controls: 500 patients without ventricular fibrillation at the acute phase of myocardial infarct.
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2007-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlation phenotype/genotype of sudden death at the acute phase of myocardial infarct. | Correlation phenotype/genotype

CONTACTS AND LOCATIONS:
Overall Officials: CHEVALIER Philippe, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital cardiologique, Lyon, France

REFERENCES:
- [Derived] Chevalier P, Roy P, Bessiere F, Morel E, Ankou B, Morgan G, Halder I, London B, Minobe WA, Slavov D, Deliniere A, Bochaton T, Paganelli F, Lesavre N, Boiteux C, Mansourati J, Maury P, Clerici G, Winum PF, Huebler SP, Carroll IA, Bristow MR. Impact of Neuroeffector Adrenergic Receptor Polymorphisms on Incident Ventricular Fibrillation During Acute Myocardial Ischemia. J Am Heart Assoc. 2023 Mar 21;12(6):e025368. doi: 10.1161/JAHA.122.025368. Epub 2023 Mar 16. PMID 36926933
- [Derived] Chevalier P, Moreau A, Bessiere F, Richard S, Chahine M, Millat G, Morel E, Paganelli F, Lesavre N, Placide L, Montestruc F, Ankou B, Puertas RD, Asatryan B, Deliniere A; MAP-IDM Investigators. Identification of Cx43 variants predisposing to ventricular fibrillation in the acute phase of ST-elevation myocardial infarction. Europace. 2023 Feb 8;25(1):101-111. doi: 10.1093/europace/euac128. PMID 35942675